CLINICAL TRIAL: NCT01102244
Title: A Study to Evaluate the Clinical Efficacy and Safety of Tobradex® ST Compared to Azasite® in the Treatment of Subjects With Moderate to Severe Chronic Blepharitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMA-09-35
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2011-01

CONDITIONS: Blepharitis
Keywords: blepharitis; moderate to severe chronic blepharitis
MeSH Terms: conditions — Blepharitis | interventions — Tobramycin, Dexamethasone Drug Combination; Azithromycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tobradex ST (Experimental): tobramycin 0.3%, dexamethasone 0.05%
  Interventions: Drug: Tobradex ST
- Azasite (Active Comparator): azithromycin 1%
  Interventions: Drug: Azasite

INTERVENTIONS:
Drug: Tobradex ST — tobramycin / dexamethasone ophthalmic suspension 0.3%/0.05% 1 drop 4 times daily for 14 days
  Arms: Tobradex ST
Drug: Azasite — azithromycin 1% 1 drop twice daily for 2 days, then once daily for 12 days
  Arms: Azasite

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of Tobradex ST compared to AzaSite in the treatment of moderate to severe chronic blepharitis.

ELIGIBILITY:
Inclusion Criteria:

* Have diagnosis of moderate to severe chronic blepharitis defined by a minimum score of at least "1" for one of the lid signs, one of the conjunctival signs, and one of the symptoms in at least one eye
* Have a minimum global score (the total signs and symptoms score) of 5 in the same eye qualifying.

Exclusion Criteria:

* Have known sensitivity or poor tolerance to the test article (tobramycin, dexamethasone, azithromycin) or its components or any therapy associated with the trial
* Have a history of ocular surgical intervention within six (6) weeks prior to Visit 1 or during the study
* Have any ocular infections (bacterial, viral or fungal) - active ocular inflammation (i.e. follicular conjunctivitis, iritis) or preauricular lymphadenopathy, other than blepharitis
* Have worn contact lenses in the 72 hours prior to visit 1 and for the duration of the study
* Are currently taking any medication known to cause ocular drying that has not been on a stable dose for at least 30 days
* Have used any topical ocular or systemic antibiotics within 7 days of enrollment. Stable (greater than 1 month prior to enrollment) use of topical antibiotics on the face (except around the eyes) for dermatologic conditions is allowed. Dose must continue unchanged for duration of study
* Have used any topical ocular - aerosolized/nebulized - or systemic corticosteroid agents within 14 days of enrollment. Stable (greater than 1 month prior to enrollment) use of inhaled (using mouthpiece) and nasal corticosteroids and topical dermal steroids (except around the eyelids) are allowed. Dose must continue unchanged for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Global sign and symptom score for blepharitis | Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- Ora, Andover, Massachusetts, United States

REFERENCES:
- [Derived] Torkildsen GL, Cockrum P, Meier E, Hammonds WM, Silverstein B, Silverstein S. Evaluation of clinical efficacy and safety of tobramycin/dexamethasone ophthalmic suspension 0.3%/0.05% compared to azithromycin ophthalmic solution 1% in the treatment of moderate to severe acute blepharitis/blepharoconjunctivitis. Curr Med Res Opin. 2011 Jan;27(1):171-8. doi: 10.1185/03007995.2010.539603. Epub 2010 Dec 7. PMID 21138337